CLINICAL TRIAL: NCT02676388
Title: Freeze-dried vs Fresh Fecal Microbiota Transplantation in Patients With Slow Transit Constipation: a Randomized Controlled Study
Brief Title: Freeze-dried vs Fresh Fecal Microbiota Transplantation in Patients With Slow Transit Constipation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, Associate professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Freeze-dried FMT-STC
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Slow Transit Constipation
Keywords: Slow Transit Constipation; Freeze-dried, Capsulized FMT; Fresh FMT
MeSH Terms: interventions — Freeze Drying

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Freeze-dried, Capsulized FMT (Experimental): Patients included will receive bowel lavage and subsequent Freeze-dried, Capsulized FMT, and then will be followed up for 3 months.
  Interventions: Procedure: Freeze-dried, Capsulized FMT
- Fresh FMT (Experimental): Patients included will receive bowel lavage and subsequent Fresh FMT, and then will be followed up for 3 months.
  Interventions: Procedure: Fresh FMT

INTERVENTIONS:
Procedure: Freeze-dried, Capsulized FMT
  Arms: Freeze-dried, Capsulized FMT
Procedure: Fresh FMT
  Arms: Fresh FMT

SUMMARY:
The purpose of this study is to compare the effect of freeze-dried, capsulized FMT and fresh FMT in adults with slow transit constipation.

DETAILED DESCRIPTION:
Constipation is a chronic disease estimated to affect about 10% - 15% of the worldwide general population. Constipation frequency appears to augment with increasing age, particularly after 65 years old.

Recent evidence in the literature and collected in the investigators' laboratory confirm that constipation can be a consequence of intestinal dysbiosis, with an increase of potentially pathogenic microorganisms and a decrease of potentially beneficial microorganisms. These alterations may affect the motility and metabolic environment of colon, especially the production of short chain fatty acids (SCFAs).

A new and under-explored method to manipulate the gastrointestinal microbiota involves fecal microbiota transplantation (FMT). There has been growing interest in the use of fecal microbiota for the treatment of patients with chronic gastrointestinal infections (e.g. CDI) and other extraintestinal conditions (e.g. IBD). Similarly, the investigators suppose that reshaping the gut microbiome with FMT would be effective for patients with slow transit constipation.

ELIGIBILITY:
Inclusion Criteria:

Chronic constipation according to Rome III criteria, defined as two or fewer spontaneous, complete bowel movements (SCBMs) per week for a minimum of 6 months;

Age ≥ 18 years;

BMI: 18.5-25 kg/m2;

Slow colonic transit confirmed by colonic transit test (colonic transit time (CTT) > 48 hours);

Normal anorectal manometry, with no evidence of dyssynergia and confirmed ability to expel rectal balloon;

No radiographic evidence of functional (i.e. pelvic floor dyssynergia) or anatomical (i.e. significant rectocele and intussusception) impediment to the expulsion of the radio-opaque contrast;

Disease duration > 1 year;

Traditional treatment with dietary modification, laxatives (including osmotic and stimulant laxatives), and biofeedback tried over the past 6 months without success;

Exclusion Criteria:

Bowel constipation due to innate factor (i.e. megacolon) or secondary interventions (i.e. drugs, endocrine, metabolic, neurologic or psychologic disorders);

History or evidence of gastrointestinal diseases (i.e. obstruction, cancer, inflammatory bowel diseases) ;

Previous abdominal surgery, except cholecystectomy, appendicectomy, tubal ligation and cesarean section;

Previous proctological or perianal surgery;

A constipation condition meeting the Rome III criteria for IBS or functional abdominal pain syndrome;

Pregnant or breast-feeding women;

Infection with enteric pathogen;

Usage of probiotics, prebiotics and/or synbiotics within the last month;

Usage of antibiotics and/or PPIs within the last 3 months;

Smoking or alcohol addiction within the last 3 months;

Uncontrolled hepatic, renal, cardiovascular, respiratory or psychiatric disease;

Disease or therapy with drugs (i.e. antidepressants, opioid narcotic analgesics, anticholinergics, calcium antagonists, nitrates, antimuscarinics) that, in the opinion of the investigator, could affect intestinal transit and microbiota.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients having on average three or more SCBMs/week | 3 months
  Proportion of patients having on average three or more spontaneous, complete bowel movements (SCBMs) per week was evaluated at week 4 and 12.

SECONDARY OUTCOMES:
Mean number of bowel movements per week | 3 months
  Patients kept daily diaries about times of bowel movements each day.
Characteristics of bowel movements | 3 months
  Patients kept daily diaries about stool consistency and degree of straining severity during defecation.
Constipation-related symptoms assessments | 3 months
  Constipation-related symptoms were evaluated using the validated Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire at week 4 and 12.
Quality-of-Life assessments | 3 months
  Quality-of-Life was evaluated using the validated Patient Assessment of Constipation Quality of Life (PAC-QOL) self-report questionnaire at week 4 and 12.
Colonic transit time measurements | 3 months
  Colonic transit time (CTT) was measured at week 4 and 12 with the Metcalf method.
Usage of laxatives or enemas as rescue medication | 3 months
  If patients did not have a bowel movement for 3 or more consecutive days, they were permitted to take up to 20 g of Macrogol 4000 powder (Forlax). If ineffective, enema was used. Patients kept daily diaries about the rescue medication when used.
Adverse events | 3 months
  Adverse events include fever, diarrhea, abdominal pain, increased bloating, borborygmi, flatulence, nausea, vomiting, nasopharyngitis, and any other disorders.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China